CLINICAL TRIAL: NCT06757348
Title: Association Between Fatty Liver and Pancreatic Steatosis in Patients With Metabolic Syndrome
Brief Title: Fatty Liver and Pancreatic Steatosis
Status: Not yet recruiting | Type: Observational
Sponsor: Maria Marta Piskorz (Other)
Responsible Party: Sponsor-Investigator, Maria Marta Piskorz, Principal Investigator, Hospital de Clinicas José de San Martín
Organization: Hospital de Clinicas José de San Martín (Other)
Other Study IDs: HCJSM-11-2024
Record Dates: First submitted 2024-10-22; First posted 2025-01-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Exocrine Pancreatic Insufficiency; Fatty Liver, Nonalcoholic; Pancreatic Steatosis
Keywords: Fatty liver; Pancreatic steatosis; Metabolic syndrome
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Non-alcoholic Fatty Liver Disease; Fatty Liver; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Fecal elastase — **Stool Samples** To investigate exocrine pancreatic insufficiency (EPI), a stool sample will be requested from all patients for fecal elastase (Fel-1) analysis. Participants will be instructed to collect their stool sample in a sterile, disposable plastic container and submit it to the Gastroenterology Chemistry Laboratory (Litwin Laboratory) for processing and analysis. Based on previously published reports, samples will be stored refrigerated at 4-8 °C for no more than 48 hours. The concentrations of Fel-1 in all samples will be measured using a commercially available enzyme-linked immunosorbent assay (ELISA) kit (ScheBo-Pancreatic Elastase 1™, Giessen, Germany), and fecal elastase will be extracted and analyzed according to the manufacturer's instructions.
Diagnostic Test: Ecoendoscopy — **Diagnosis of Pancreatic Steatosis** The diagnosis of pancreatic steatosis will be performed using endoscopic ultrasound. A Pentax EG-3870UTK endoscope will be used in conjunction with Hitachi Avius ultrasound equipment. The procedure is performed under anesthesia using propofol.
Diagnostic Test: Fibroscan — **Fibroscan Procedure:** This is a new technique based on the evaluation of liver elasticity or stiffness that allows for the measurement of liver hardness and quantification of liver fibrosis in a simple and completely painless manner using ultrasound. The results are obtained immediately and can be safely repeated periodically.
Diagnostic Test: Serum cytokines — Peripheral blood will be drawn from all participants in the Gastroenterology Division of the Hospital de Clínicas. Samples will be collected in EDTA tubes, centrifuged, and the serum will be frozen at -80 °C until processing. Serum cytokine levels will be measured using a commercial kit (Bio-Plex Pro human cytokine, Bio-Rad Lab., Inc.), which includes a panel of 27 cytokines: FGF basic, Eotaxin, G-CSF, GM-CSF, IFN-γ, IL-1β, IL-1ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, MIP-1α, IL-12 (p70), MIP-1β, IL-13, PDGF-BB, IL-15, RANTES, IL-17, TNF-α, IP-10, VEGF, MCP-1 (MCAF).

SUMMARY:
The goal of this observational study is to determine the prevalence of pancreatic steatosis in patients with fatty liver and determine the prevalence of exocrine pancreatic insufficiency (EPI) in these patients.

Participants with fatty liver and metabolic syndrome will undergo fecal elastase measurement and endoscopic ultrasound (EUS).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the association between non-alcoholic fatty liver disease and non-alcoholic pancreatic steatosis and to describe cytokine levels in the context of a global epidemic of obesity and metabolic syndrome, which could represent a new treatment target in previously underdiagnosed patients with pancreatic insufficiency and pancreatic steatosis.

Patients over 18 years old with a diagnosis of MAFLD (Metabolic Dysfunction-Associated Fatty Liver Disease) will undergo the following assessments:

* Exocrine Pancreatic Insufficiency Questionnaire (PEI-Q)
* Measurement of weight, height, and abdominal circumference
* Fecal elastase (Fel-1)
* Pro-inflammatory and anti-inflammatory cytokines in serum
* Hydrogen and methane breath tests to evaluate small intestinal bacterial overgrowth (SIBO)
* Endoscopic ultrasound with sedation
* Fibroscan Exocrine pancreatic insufficiency (EPI) will be defined as a fecal elastase-1 (Fel-1) concentration of < 100 µg/g or Fel-1 between 100 and 200 µg/g with alterations in additional pancreatic pathology tests, such as serum albumin, vitamin E, vitamin D, vitamin A, folic acid, iron, transferrin, calcium, magnesium, and/or malnutrition identified through anthropometric measurements conducted by an expert nutritionist. Fel-1 ≥ 200 µg/g will be considered normal.

Additionally, for those patients with fecal elastase levels below 200 µg/g, the following measurements will be conducted:

* Proteinogram
* Vitamin E, vitamin D, vitamin A, vitamin K
* Folic acid, B12
* Calcium, magnesium, zinc
* Iron profile
* Nutritional assessment with anthropometry

For those with exocrine pancreatic insufficiency (EPI):

* IgG4
* Alpha-1 antitrypsin
* Endoscopic ultrasound (EUS) with biopsies

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with a diagnosis of Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD).

Exclusion Criteria:

* - Alcohol consumption >20 g/day in women, >30 g/day in men
* Chronic hepatitis B or C infection
* Autoimmune liver diseases: autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis
* Hereditary hemochromatosis
* Wilson's disease
* Alpha-1 antitrypsin deficiency
* Celiac disease
* Uncontrolled thyroid disease
* Active or chronic infectious disease
* Active cancer or ongoing treatment
* Chronic renal insufficiency
* Pregnancy/lactation
* Insufficient data
* Patients who do not complete follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with a diagnosis of Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD).
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence Non-Alcoholic Fatty Pancreas Disease | At baseline
  Determine the prevalence of Non-Alcoholic Fatty Pancreas Disease (NAFPD) in patients with Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD).
Prevalence of exocrine pancreatic insufficiency | At baseline
  Determine the prevalence of exocrine pancreatic insufficiency (EPI) in patients with Non-Alcoholic Fatty Pancreas Disease (NAFPD).
Prevalence of IPE in MAFLD | At baseline
  Determine the prevalence of exocrine pancreatic insufficiency (EPI) in patients with Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD).

SECONDARY OUTCOMES:
Clinical characteristics | At baseline
  Analyze the causes of exocrine pancreatic insufficiency (EPI) and Non-Alcoholic Fatty Pancreas Disease (NAFPD) in this population.
Cytokine profile | At baseline
  Evaluate the cytokine phenotypic profile in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clinicas Jose de San Martin, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
The data sets, including the redacted study protocol, redacted statistical analysis plan, and individual participant data supporting the results reported in this article, will be made available within 3 months from initial request to researchers who provide a methodologically sound proposal. The data will be provided after its de-identification, in compliance with applicable privacy laws, data protection, and requirements for consent and anonymization.

REFERENCES:
- [Result] Olmos JI, Piskorz MM, Litwin N, Schaab S, Tevez A, Bravo-Velez G, Uehara T, Hashimoto H, Rey E, Sorda JA, Olmos JA. Exocrine Pancreatic Insufficiency is Undiagnosed in Some Patients with Diarrhea-Predominant Irritable Bowel Syndrome Using the Rome IV Criteria. Dig Dis Sci. 2022 Dec;67(12):5666-5675. doi: 10.1007/s10620-022-07568-8. Epub 2022 Jun 15. PMID 35704255
- [Result] Bellentani S. The epidemiology of non-alcoholic fatty liver disease. Liver Int. 2017 Jan;37 Suppl 1:81-84. doi: 10.1111/liv.13299. PMID 28052624
- [Result] Bedogni G, Miglioli L, Masutti F, Castiglione A, Croce LS, Tiribelli C, Bellentani S. Incidence and natural course of fatty liver in the general population: the Dionysos study. Hepatology. 2007 Nov;46(5):1387-91. doi: 10.1002/hep.21827. PMID 17685472
- [Result] Weiss J, Rau M, Geier A. Non-alcoholic fatty liver disease: epidemiology, clinical course, investigation, and treatment. Dtsch Arztebl Int. 2014 Jun 27;111(26):447-52. doi: 10.3238/arztebl.2014.0447. PMID 25019921
- [Result] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314
- [Result] Eslam M, Newsome PN, Sarin SK, Anstee QM, Targher G, Romero-Gomez M, Zelber-Sagi S, Wai-Sun Wong V, Dufour JF, Schattenberg JM, Kawaguchi T, Arrese M, Valenti L, Shiha G, Tiribelli C, Yki-Jarvinen H, Fan JG, Gronbaek H, Yilmaz Y, Cortez-Pinto H, Oliveira CP, Bedossa P, Adams LA, Zheng MH, Fouad Y, Chan WK, Mendez-Sanchez N, Ahn SH, Castera L, Bugianesi E, Ratziu V, George J. A new definition for metabolic dysfunction-associated fatty liver disease: An international expert consensus statement. J Hepatol. 2020 Jul;73(1):202-209. doi: 10.1016/j.jhep.2020.03.039. Epub 2020 Apr 8. PMID 32278004
- [Result] Dominguez-Munoz JE. Diagnosis and treatment of pancreatic exocrine insufficiency. Curr Opin Gastroenterol. 2018 Sep;34(5):349-354. doi: 10.1097/MOG.0000000000000459. PMID 29889111